CLINICAL TRIAL: NCT00712257
Title: A Prospective, Multicenter Trial to Evaluate the Safety and Performance of Spectranetics Laser With Adjunct PTA and GORE VIABAHN Endoprosthesis for the Treatment of SFA Instent Restenosis.
Brief Title: Study to Evaluate the Safety and Performance of Spectranetics Laser w/Adjunct PTA and Gore Viabahn Endoprosthesis for Treatment of SFA Instent Restenosis
Acronym: SALVAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to safety concerns
Sponsor: VIVA Physicians (Other)
Collaborators: W.L.Gore & Associates (Industry); Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SALVAGE - 00106-661
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Restenosis
Keywords: treatment of superficial femoral artery instent restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spectranetics Laser plus Gore Viabahn Endoprosthesis (Other): Spectranetics Laser for optimal debulking followed by adjunctive PTA plus GORE VIABAHN Endoprosthesis with Heparin Bioactive Surface placement
  Interventions: Device: Spectranetics Laser with adjunct PTA and Gore VIABAHN Endoprosthesis with Heparin Bioactive Surface

INTERVENTIONS:
Device: Spectranetics Laser with adjunct PTA and Gore VIABAHN Endoprosthesis with Heparin Bioactive Surface — treatment for superficial femoral artery instent re-stenosis

SUMMARY:
A Multicenter study to evaluation the safety and performance of Spectranetics Laser with Adjunct PTA and Gore Viabahn Endoprosthesis for the Treatment of SFA Instent Restenosis

ELIGIBILITY:
Inclusion Criteria:

* Subject or subject's legal representative informed of the study nature.
* Subject understands the duration of the study and its follow up visit requirements.
* Intermittent claudication extending through critical limb ischemia meeting a Rutherford 2-5 category.
* Subject able to walk unassisted.
* Female subjects of childbearing potential must have a negative serum pregnancy test 7 days prior to treatment.

Exclusion Criteria:

* Life expectancy less than 12 months
* Myocardial infarction less than 3 months prior to procedure
* Known allergies or sensitivities to heparin, aspirin, other anti-coagulant/antiplatelet therapies and nitinol.
* Known allergy to contrast media that cannot adequately be pre-medicated prior to study procedure.
* Uncontrolled hypercoagulability

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
12-month duplex-ultrasound defined target lesion patency will be assessed in the enrollment arm. Patency is defined as a ratio of less than 2.0, measured as the upstream peak systolic velocity compared with PSV in the area of greatest stenosis. | 12 months

SECONDARY OUTCOMES:
Target lesion revascularization will be evaluated at 12 mos. and defined as any pecutaneous or surgical intervention to treat a stenosis or cocclusion of the arget lesion treated at the index procedure. | 12 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Tony Das, MD, Principal Investigator — Presbyterian Heart Institute
Locations (1):
- Gary Ansel, MD, Columbus, Ohio, United States